CLINICAL TRIAL: NCT02237391
Title: Evaluation of a Complex Interdisciplinary Pain Assessment Program Linked to Primary Care to Improve Clinical Outcomes and Reduce Health Care Utilization Among Patients With Chronic Pain and Frequent Emergency Department Visits
Brief Title: Evaluation of a Interdisciplinary Pain Program Among Patients With Chronic Pain and Frequent Emergency Department Visits
Acronym: CIPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20140575-01H
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain; Peer Review, Health Care; Interdisciplinary Communication
Keywords: High Frequency Emergency Department Visits; Healthcare Utilization; Chronic Pain; Interdisciplinary
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIPAP Program (Experimental): Complex Interdisciplinary Pain Assessment Program
  Interventions: Other: CIPAP Program
- Treatment as Usual (TAU) (Other): Treatment as usual control group
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: CIPAP Program — The intervention will involve a pain specialist, a clinical health psychologist and a nurse. As needed, it may involve a social worker, an addiction specialist, and other specialists. The pain specialist will conduct an evaluation that includes: history of presenting illness, review of systems, review of pain treatments, medical history, surgical history, addiction history, medications and allergies, insurance for medication, psychosocial history, opioid risk assessment, physical examination, and review of tests and investigations. The psychologist will conduct an evaluation that includes: a structured diagnostic clinical interview, a review of coping strategies, and a review of the questionnaires completed prior to the assessment pertaining to mood, anxiety, trauma and beliefs about pain.
  Other Names: Complex Interdisciplinary Pain Assessment Program
  Arms: CIPAP Program
Other: Treatment as Usual (TAU) — Control group
  Other Names: Treatment as Usual control group
  Arms: Treatment as Usual (TAU)

SUMMARY:
While significant advances in pain management have occurred in the last 20 years, the majority of patients with chronic pain (CP) are unable to access evidence-based treatment at either the primary or tertiary care level.

Moreover, research has shown that unrelieved CP and the lack of available expertise contribute to emergency department (ED) visits and hospital admissions. At The Ottawa Hospital (TOH), close to 18,000 ED visits per year are related to CP (12.9%). Among high frequency visitors (HFV; >= 8 visits per year), a small number of patients with CP use an inordinate amount of acute care resources. The investigators study will use a randomized controlled (RCT) design to conduct a pilot evaluation of the impact of a Complex Interdisciplinary Pain Assessment Program (CIPAP) linked with primary care physicians (PCP) compared to a treatment as usual (TAU) control arm.

The investigators hypothesis is that implementing a CIPAP will increase health care value through improved patient outcomes and reduced costs in HFV with chronic pain (CP-HFV). The investigators believe that a CIPAP will provide CP-HFV patients long-term pain management solutions, ED visits for CP will be reduced, and hospital admissions for CP will be prevented. This pilot RCT study will inform a larger-scale RCT study to be conducted in the future.

DETAILED DESCRIPTION:
As this is a phase 2 trial, the sample size is primarily determined by logistical constraints; however, as this trial will yield valuable information about the preliminary impact of the program for planning a larger, more definitive trial in the future, we determined the maximum width of a two-sided 95% confidence interval around the differences between the arms at 12 months. For self-report measures, 18 patients per arm would yield a margin of error of 0.65 standard deviations (total width of confidence interval = 1.3 on the standard deviation unit scale), which is considered acceptable for the self-report measures. For number of visits over 3 months, we assumed a standard deviation of 3 (based on our preliminary data). Assuming approximate normality, our sample size of 18 patients per arm would yield a margin of error of 2 visits (total width of confidence interval = 4 visits) which is adequate to yield preliminary evidence of change. These are conservative estimates as our analyses will include repeated measures, and adjust for baseline measures of response in addition to other demographic and clinical covariates. To account for 20% attrition, we will plan to enrol 23 participants per arm (total number of participants =46).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years old)
* Working knowledge of English or French
* Presented to The Ottawa Hospital Emergency Department (TOH ED) with a primary complaint of chronic or recurrent pain a minimum of 8 times over the last 12 months, with 3 of the visits occurring in the 3 months prior to study enrollment.
* Patients fit criteria for chronic pain (CP) if they have had "pain that has lasted longer than three months." As per the International Association for the Study of Pain (IASP) taxonomy of CP syndromes, this includes: "relatively generalized syndromes," "relatively localized syndromes of the head and neck," "spine and radicular pain syndromes," "local syndromes of the upper limbs," and "visceral pain syndromes."

Exclusion Criteria:

* Malignant pain - patients will be referred to our complex cancer pain program
* Canadian Triage and Acuity Scale Level 1 and Level 2; Level 3 will be assessed on a case-by-case basis and we will document reason for exclusion
* Refusal or inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-12; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  The primary outcome is pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale. The Brief Pain Inventory (BPI) - Pain Interference consists of 7 numerical scales (0 to 10) rating pain interference with general activity, mood, walking ability, work, relations with other people, sleep and enjoyment of life.

SECONDARY OUTCOMES:
Change from baseline in pain catastrophizing, as measured by the Pain Catastrophizing Scale, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  Pain Catastrophizing Scale (PCS): The PCS is a 13-item self-report measure that uses a 5-point Likert scale allowing participants to rate the degree to which they adopt a negative or aversive orientation towards their pain. The PCS has a stable three-factor structure (rumination, magnification, and helplessness).
Change from baseline in self-reported anxiety, as measured by the Generalized Anxiety Disorder Scale - 7, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  Generalized Anxiety Disorder Scale-7 (GAD-7): The GAD-7 will be used to evaluate symptoms of anxiety. It is a 7-item self-report measure that uses a 4-point Likert scale allowing participants to rate themselves with scores of either 0,1,2 or 3 (representing answers of "not at all," "several days," "more than half the days," and "nearly every day," respectively). Total scores range from 0-21 with cut-off points of 5, 10 and 15 representing mild, moderate and severe anxiety, respectively.
Change from baseline in self-reported depressive symptoms, as measured by the Patient Health Questionnaire - 9, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  Patient Health Questionnaire-9 (PHQ-9): The PHQ-9 will be used to evaluate depressive symptoms. This 9-item scale assesses the frequency of depressive symptoms experienced over the past two weeks.
Change from baseline in self-reported sleep problems, as measured by the Insomnia Severity Index, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  Insomnia Severity Index (ISI): The ISI is a 7-item self-report questionnaire that evaluates the severity of initial insomnia, sleep maintenance problems, terminal insomnia, satisfaction with sleep patterns, interference with daily functioning, impairment attributed to sleep problems and level of distress caused by sleep problems. It uses a 5-point Likert scale (0 = not at all; 4 = extremely), total scores range from 0 to 28, with high scores indicating greater insomnia severity.
Change from baseline in risk for opioid abuse, as measured by the Screener and Opioid Assessment for Patients with Pain, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  Screener and Opioid Assessment for Patients with Pain (SOAPP): The SOAPP is a 24-item questionnaire used to evaluate the risk for opioid abuse in patients with chronic pain who are being considered for long-term opioid therapy. A consensus of 26 pain and addiction experts was obtained in order to determine the important characteristics of patients with chronic pain that can predict medication misuse. Fourteen of the 24 SOAPP items predict future aberrancies.
Change from baseline in self-reported traumatic stress, as measured by the PTSD Checklist for DSM - 5, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  PTSD Checklist for DSM - 5 (PCL-5): The PCL-5 is a self-report questionnaire that assesses symptoms for post-traumatic stress disorder (PTSD). It is used as a measure of the 20 symptoms of PTSD that are mentioned in the Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-V) and has been validated. Each item on the questionnaire is rated on a scale of 0 to 4, representing answers of "not at all," "a little bit," "moderately," "quite a bit," and "extremely," respectively. Total scores range from 0-80 with a cut-off point of 38 suggesting endorsement of PTSD.
Change from baseline in self-reported quality of life, as measured by The Quality of Life Questionnaire EuroQol, at 12-months post-study enrollment | Baseline and 12 months post-enrollment
  The Quality of Life Questionnaire EuroQol (EQ-5D): The EQ-5D is a simple-to-use, valid, and sensitive instrument measuring quality of life. It covers 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, or severe problems and participants use a tick box to select the statement that is most representative of their conditions. Participants are also asked to rate, using a visual analogue scale (0 to 100), their state of health.
Change from 3-months pre-study enrollment in healthcare utilization, as measured by the Pain Economics Questionnaire, at 12-months post-study enrollment | 3 months pre-study and 12 months post-enrollment
  The Pain Economics Questionnaire (PEQ): The PEQ is a brief self-report questionnaire created for this study to obtain information regarding participants' health care utilization. This questionnaire has not been tested for reliability or validity. It will be used to capture participants' use of non-The Ottawa Hospital Emergency Department (TOH ED) hospitalizations, family doctor visits, diagnostic tests, surgeries, allied health care visits and medications.
Change from 3-months pre-study enrollment in healthcare utilization, as measured by participant Ministry of Health and Long-Term Care Personal Claims History Information, at 12-months post-study enrollment | 3 months pre-study and 12 months post-enrollment
  With participant consent, we will be requesting information regarding participants' health care utilization from Ministry of Health and Long-Term Care (MOHLTC).
Change from 3-months pre-study enrollment in opioid usage, as measured by morphine equivalents, at 12-months post-study enrollment | 3 months pre-study and 12 months post-enrollment
  With participant consent, we will be requesting medication information from participants' pharmacy and calculating morphine equivalent values for all opioids prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Smyth, MD PhD, Principal Investigator — Ottawa Hospital Research Institute; Patricia Poulin, PhD C.Psych, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No